CLINICAL TRIAL: NCT02594878
Title: Chronic Non-bacterial Osteomyelitis Treated With Pamidronate in a Randomised Placebo Controlled Trial
Brief Title: Chronic Non-bacterial Osteomyelitis Treated With Pamidronate
Acronym: CNOPAM
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 48438
Record Dates: First submitted 2015-10-20; First posted 2015-11-03 (Estimated); Last update posted 2016-11-16 (Estimated); Status verified 2016-11

CONDITIONS: Immune System Disease; Musculoskeletal Disease
Keywords: Chronic non-bacterial osteomyelitis; Chronic recurrent multifocal osteomyelitis; Non- bacterial osteomyelitis; SAPHO syndrome; Whole body MRI; Pamidronate; Inflammatory bone disease; Autoinflammatory disease
MeSH Terms: conditions — Immune System Diseases; Musculoskeletal Diseases; Chronic recurrent multifocal osteomyelitis; Acquired Hyperostosis Syndrome; Osteitis | interventions — Pamidronate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pamidronatdinatrium 3mg/ml (Experimental): Pamidronatdinatrium 1 mg/kg max 60 mg for 3 days every 3 month in total of 3 series (0,3,6 month). First day first series 0,5mg/kg max 30 mg.
  Interventions: Drug: Pamidronatdinatrium
- Natrium chloride 9 mg/ml (Placebo Comparator): Natrium chloride 9 mg/ml volume equals experimental drug
  Interventions: Other: Natrium chloride 9mg/ml

INTERVENTIONS:
Drug: Pamidronatdinatrium
  Other Names: Pamidronat, Pamifos, Aredia
  Arms: Pamidronatdinatrium 3mg/ml
Other: Natrium chloride 9mg/ml
  Arms: Natrium chloride 9 mg/ml

SUMMARY:
In a randomized double blind placebo controlled trial to investigate the effect of pamidronate in treatment of chronic non bacterial osteomyelitis.

Main objective:

1. Reduction of the inflammatory activity in the bone lesions measured by whole body MRI after 36 weeks.
2. Healing of the inflammatory activity in the bone lesions measured by whole body MRI after 36 weeks.

Secondary objectives:

1. Changes in bone lesions in whole body MRI between baseline and week 12 and between week 12 and week 36
2. Changes in bone lesions of anterior chest-wall (adults) evaluated by CT scan between baseline and week 36.
3. Changes in patient self reported outcome measures
4. Changes in inflammatory markers and bone markers.

DETAILED DESCRIPTION:
Chronic non-bacterial osteomyelitis is a multifocal inflammatory bone disorder. The pathogenesis is unknown. The disease is mainly diagnosed in childhood. There is a strong association with inflammatory disorders of the skin, mainly psoriasis. The disease is characterized by recurrent episodes of pain and disability. It is unclear if SAPHO syndrome (synovitis, acne, pustulosis, hyperostosis, osteitis) might be the adult version of chronic non-bacterial osteomyelitis. The disease can persist in adulthood and course chronic bone deformations.

Wholebody MRI is the most sensitive imaging for diagnosing and monitoring the non bacterial osteitis.

The treatment of chronic non-bacterial osteomyelitis is largely empiric. First line treatment is NSAID (Non Steroidal Anti-Inflammatory Drug). When NSAID is inadequate the bisphosphonate pamidronate has been described relief pain in small cohorts in retrospective studies.

In this research protocol, investigators seek to investigate if it is beneficial to use pamidronate in the treatment of chronic non bacterial osteomyelitis and the osteitis component in SAPHO syndrome. Primary outcome is whole body MRI. Secondary outcome is CT scan, patient measure reported outcome and biomarkers. A biobank may help us to understand the pathogenesis and future treatment targets of chronic non bacterial osteomyelitis.

ELIGIBILITY:
Inclusion Criteria:

* Age: 9-65 years (inclusive)
* Fulfilling the diagnostic criteria for chronic non bacterial osteomyelitis:

  1. Mono-, oligo- or multifocal inflammatory bone lesions (osteomyelitis, osteitis, osteosclerosis)
  2. Diagnostic score according to A. Jansson criteria (2009) > 39 or malignancy and infection excluded by biopsy
  3. Symptoms > 6 weeks
* Volunteer, signed written informed content

Exclusion Criteria:

* Age older than 65 years
* Age younger than 9 years
* Pregnant women or nursing (breastfeeding) mothers
* Hypersensitivity to pamidronate, bisphosphonate og additives in pamidronate
* Known history or current lymphoproliferative disease
* History of surgery on glandula thyroidea
* Known alcohol/medical abuse
* Poor dental status
* Low Vitamin D- status
* Liver/ kidney disease
* Abnormal laboratory screening for comorbidity

Ages: 9 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2015-10; Primary Completion 2018-05 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Wholebody MRI | Changes between baseline and week 36

SECONDARY OUTCOMES:
CT scan of the anterior chestwall (adults) | Changes between baseline and week 36
Systemic inflammatory markers | Changes between baseline and week 1, 4, 12, 24 and 36
  TNF- α,IL-1 β, IL-8, IL-18, IL-17, INF-ƴ, IL-6, IL-10, IL-11, IL-21, MIP 1-alfa (CCL3, 22) and IL-1Ra
Systemic bone markers | Changes between baseline and week 1, 4, 12, 24 and 36
  s-CTX og s-NTX, P1NP, C1NP, TRACP 5b, bone alkaline phosphatase
Wholebody MRI | Changes between baseline and week 12 and changes between week 12 and 36
Changes in Health Assesment Questionnaire score | Changes between baseline and week 1, 4, 12, 24 and 36
Changes in Children Assesment Questionnaire score | Changes between baseline and week 1, 4, 12, 24 and 36
Changes in Visual Analog Score for pain | Changes between baseline and week 1, 4, 12, 24 and 36

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Marie Andreasen, MD, Principal Investigator — University hospital of Aarhus, Denmark
Locations (1):
- Universityhospital of Aarhus, Denmark, Aarhus, Denmark

REFERENCES:
- [Derived] Andreasen CM, Jurik AG, Deleuran BW, Horn HC, Folkmar TB, Herlin T, Hauge EM. Pamidronate in chronic non-bacterial osteomyelitis: a randomized, double-blinded, placebo-controlled pilot trial. Scand J Rheumatol. 2020 Jul;49(4):312-322. doi: 10.1080/03009742.2020.1724324. Epub 2020 Jun 2. PMID 32484386